CLINICAL TRIAL: NCT03471247
Title: CYCLE RCT: An International, Multi-centre, Randomized Clinical Trial of Early In-bed Cycling for Mechanically Ventilated Patients
Brief Title: CYCLE: A Randomized Clinical Trial of Early In-bed Cycling for Mechanically Ventilated Patients
Acronym: CYCLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Critical Care Trials Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYCLE RCT
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Intensive Care Unit Acquired Weakness; Critical Care; Mechanical Ventilation; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Bed Cycle Ergometer + Routine PT (Experimental): Patients will receive 30 minutes of in-bed cycling once per day, 5 days per week, while they remain in the ICU, for up to a maximum of 28 days. They will also receive routine physiotherapy.
  Interventions: Device: In-Bed Cycle Ergometer; Other: Routine PT
- Routine PT (Active Comparator): Patients will receive routine physiotherapy interventions per current institutional practice
  Interventions: Other: Routine PT

INTERVENTIONS:
Device: In-Bed Cycle Ergometer — Physiotherapists will place the patient's legs in a specialized in-bed cycle ergometer allowing for gentle leg exercise. Exercise can performed in passive, active-assisted, or active mode.
  Other Names: Restorative Therapies RT300 Supine
  Arms: In-Bed Cycle Ergometer + Routine PT
Other: Routine PT — Includes, based on the patient's alertness and medical stability, activities to maintain or increase limb range of motion and strength, in- and out- of bed mobility, ambulation, and assistance with optimizing airway clearance and respiratory function.

SUMMARY:
Patients who survive critical illness usually experience long-lasting physical and psychological impairments, which are often debilitating. Rehabilitation interventions started in the ICU may reduce this morbidity. In-bed cycling, which uses a special bicycle that attaches to the hospital bed, allows critically ill patients who are mechanically ventilated (MV) to gently exercise their legs while in the ICU. The main goal of this study is to determine whether critically ill MV adults recover faster if they receive early in-bed cycling than if they do not. Another objective is to determine whether in-bed cycling is a cost-effective intervention. 360 patients admitted to the ICU and receiving MV will be enrolled in the study. Following informed consent, patients will be randomized to either (1) early in-bed cycling and routine physiotherapy or (2) routine physiotherapy alone. Patients' strength and physical function will be measured throughout the study. If early in-bed cycling during critical illness improves short-term physical and functional outcomes, it could accelerate recovery and reduce long-term disability in ICU survivors.

DETAILED DESCRIPTION:
Background: Survivors of critical illness have a long road of physical, cognitive, and psychological recovery. Although medical advances have reduced the mortality of critical illness, survival often comes with substantial long-term morbidity and societal cost. At 1-year follow-up, ~35% of intensive care unit (ICU) survivors had sub-normal 6-minute walk distance, and ~50% had not returned to work. Rehabilitation interventions started in the ICU may reduce this morbidity. In-bed cycling is a novel technology that may help critically ill, mechanically ventilated (MV) patients receive exercise very early to prevent or attenuate muscle weakness. Patients on MV typically receive prolonged bedrest and are often perceived as 'too sick' for physiotherapy (PT) interventions. However expert consensus and our previous multicentre pilot work suggest these interventions are safe. The CYCLE RCT will evaluate whether early in-bed cycling compared to usual PT interventions improves patient-reported outcomes.

Objectives:

1. CYCLE RCT: To determine if early in-bed cycling and routine PT compared to routine PT alone in critically ill, mechanically ventilated adults improves the primary outcome of physical function at 3 days after ICU discharge and secondary outcomes of strength, physical function, frailty, psychological distress, quality of life, mortality, and healthcare utilization.
2. Economic Evaluation: To determine the cost-effectiveness of cycling and routine PT compared to routine PT alone among critically ill, mechanically ventilated adults.

Design: 360-patient concealed open-label RCT with blinded outcome assessment

Population: Critically ill adults receiving MV in a medical-surgical ICU

Methods: After informed consent, patients will be randomized to receive 30 minutes/day of cycling, 5 days per week and routine PT interventions or routine PT interventions alone. Assessors, blinded to treatment allocation, will measure the primary outcome of patients' physical function at 3 days post-ICU. Secondary outcomes will be measured at ICU awakening, ICU discharge, 3 days post-ICU, hospital discharge, and 90-days post-enrollment.

Relevance: By 2026, demand for ICU services is estimated to increase by 40% and more survivors will be at risk for post-ICU disability. If early cycling during critical illness improves short-term physical and functional outcomes, it could accelerate recovery and reduce long-term disability in ICU survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age
* Patient is invasively mechanically ventilated ≤ 4 days
* Expected additional 2 day ICU stay
* Ability to ambulate independently (with or without gait aid) before their critical illness
* ICU length of stay ≤ 7 days

Exclusion Criteria:

* Pre-hospital inability to follow simple commands in local language at baseline
* Acute conditions impairing ability to receive cycling
* Severe cognitive impairment pre-ICU
* Traumatic brain injury
* Acute proven or suspected central or peripheral neuromuscular weakness affecting the legs (e.g., stroke, Guillian-Barre syndrome, spinal injury)
* Temporary pacemaker (internal or external)
* Expected hospital mortality ≥ 90%
* Equipment unable to fit patient's body dimensions (elg., leg amputation, morbid obesity)
* Palliative goals of care
* Pregnancy (suspected or proven)
* Specific surgical exclusion as stipulated by surgery or ICU team
* Physician declines
* Cycling exemption not resolved during first 4 days of mechanical ventilation
* Patient already able to march on spot at time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Physical Function Test for ICU-scored (PFIT-s) | 3 days after ICU discharge
  Patients complete 4 activities: arm and leg strength, ability to stand, and step cadence. Scores range from 0 to 10, with higher scores = better function.

SECONDARY OUTCOMES:
Physical Function Test for ICU-scored (PFIT-s) | ICU Awakening, approximately 6 days after ICU admission; ICU Discharge, approximately 12 days after ICU admission; Hospital Discharge, approximately 28 days after ICU admission
  Patients complete 4 activities: arm and leg strength, ability to stand, and step cadence. Scores range from 0 to 10, with higher scores = better function.
Muscle Strength | ICU Awakening, approximately 6 days after ICU admission; ICU Discharge, approximately 12 days after ICU admission; 3 days after ICU discharge; Hospital Discharge, approximately 28 days after ICU admission
  Manual muscle testing using the Medical Research Council (MRC) Scale. The patient exerts a force against the examiner's resistance. Each muscle is assessed on a 6-point scale (0 = no contraction, 5 = contraction sustained against maximal resistance). Scores range from 0 to 60, with higher scores = better strength.
30 Second Sit to Stand | ICU Awakening, approximately 6 days after ICU admission; ICU Discharge, approximately 12 days after ICU admission; 3 days after ICU discharge; Hospital Discharge, approximately 28 days after ICU admission
  Patient completes as many sit to stand repetitions as possible in 30 seconds. Total number of repetitions is recorded as patient's score. Higher repetitions represent better function.
Two Minute Walk Test | ICU Discharge, approximately 12 days after ICU admission; 3 days after ICU discharge; Hospital Discharge, approximately 28 days after ICU admission
  Maximum distance walked in 2 minutes measured in metres on a continuous scale.
Patient-Reported Functional Scale-ICU (PRFS-ICU) | ICU discharge, approximately 12 days after ICU admission; hospital discharge, approximately 28 days after ICU admission; 3 months after enrollment
  Assesses patient's perception of their physical function. Patients rate their ability to perform 6 mobility activities on a 0-10 scale (0=unable to perform activity, 10=able to perform activity at same level as before ICU admission). Scores range from 0 to 60, with higher scores representing better function.
Katz Activities of Daily Living (ADL) Scale | Baseline; ICU discharge, approximately 12 days after ICU admission; hospital discharge, approximately 28 days after ICU admission
  Rates the patient's ability to complete 6 tasks: bathing, dressing, toileting, feeding, continence, and bed mobility. A rater assesses whether the patient is dependent or independent according to pre-specified criteria. Scores range from 0 to 6, with higher scores representing better function.
Clinical Frailty Scale | Baseline; hospital discharge, approximately 28 days after ICU admission
  Patients are ranked on a scale from 1-9 according to level of frailty based on clinical descriptions (1 = very fit, 9 = terminally ill).
Intensive Care Psychological Assessment Tool (IPAT) | After ICU awakening assessment, approximately 7 days after ICU admission
  Patients answer 10 questions related to critical care-related psychological distress. Scores range from 0-20, with scores of 7 or greater indicating a patient at risk of future psychological morbidity.
Duration of Mechanical Ventilation | From study admission to ICU discharge, approximately 10 days
  Duration of invasive mechanical ventilation
Length of stay | From hospital admission to ICU discharge (approximately 14 days) and hospital discharge (approximately 21 days)
  ICU and Hospital length of stay
Health-Related Quality of Life - EuroQol-5D-5L and Visual Analogue Scale | ICU discharge, approximately 12 days after ICU admission; hospital discharge, approximately 28 days after ICU admission; 3 months after enrollment
  Five question self-administered, preference-based instrument to measure mobility, self-care, usual activities, pain, and anxiety/depression, as well as a visual analogue scale (VAS) global assessment of health. For each dimension, the participant chooses 1 of 5 levels that best describes their health on that day: "no problem" (1), "slight" (2), "moderate" (3), "severe" (4), or "unable/extreme" (5). The VAS is the participant's rating of their health on a scale of 0 "worst health you can imagine" to 100 "best health you can imagine".
Mortality | From study admission to 3 months after enrollment
  Death in ICU, hospital, or post-discharge.
Hospital Discharge Location | Hospital discharge, approximately 28 days after ICU admission
  For survivors: home, inpatient rehabilitation, other hospital, chronic care, assisted living facility, nursing home.
Hospital Anxiety and Depression Scale (HADS) | 3 months after enrollment
  Patient answers 14 questions related to anxiety and depression. Scores range from 0-21 with higher score indicating more distress.
Quality-Adjusted Life Years (QALYs) | 3 months after enrollment
  A measure of health outcomes for economic evaluation that incorporates the impact of an intervention on both the quantity and quality of life.
Healthcare Utilization | From study admission to 3 months after enrollment
  Includes emergency room visits and hospitalizations, family doctor visits, specialist visits and outpatient clinics, other healthcare professional services.
Intervention and Healthcare Costs | From study admission to 3 months after enrollment
  Includes emergency room visits and hospitalizations, family doctor visits, specialist visits and outpatient clinics, assistive devices, renovations and modifications, other healthcare professional services, employment status and time off work, assistance from others.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kho, PT, PhD, Principal Investigator — McMaster University School of Rehabilitation Science
Locations (16):
- United States (2):
  - University of Maryland Medical Centre, Baltimore, Maryland
  - Duke University Hospital, Durham, North Carolina
- Austin Health - Austin Hospital, Heidelberg, Victoria, Australia
- Canada (13):
  - Brant Community Healthcare System - Brantford General Hospital, Brantford, Ontario
  - Hamilton Health Sciences - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences - Juravinski Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Niagara Health System - St. Catharines Site, St. Catharines, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Centre Integre de Sante et de Services Sociaux de Chaudiere-Appalaches - Hotel-Dieu de Levis, Lévis, Quebec
  - Centre Integre Universitaire de Sante et de Services Sociaux du Nord-de-L'Ile-de-Montreal - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - Centre Integre Universitaire de Sante et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid JC, Molloy A, Strong G, Kelly L, O'Grady H, Cook D, Archambault PM, Ball I, Berney S, Burns KEA, D'Aragon F, Duan E, English SW, Lamontagne F, Pastva AM, Rochwerg B, Seely AJE, Serri K, Tsang JLY, Verceles AC, Reeve B, Fox-Robichaud A, Muscedere J, Herridge M, Thabane L, Kho ME; CYCLE Investigators. Research interrupted: applying the CONSERVE 2021 Statement to a randomized trial of rehabilitation during critical illness affected by the COVID-19 pandemic. Trials. 2022 Sep 2;23(1):735. doi: 10.1186/s13063-022-06640-y. PMID 36056378
- [Background] Kho ME, Reid J, Molloy AJ, Herridge MS, Seely AJ, Rudkowski JC, Buckingham L, Heels-Ansdell D, Karachi T, Fox-Robichaud A, Ball IM, Burns KEA, Pellizzari JR, Farley C, Berney S, Pastva AM, Rochwerg B, D'Aragon F, Lamontagne F, Duan EH, Tsang JLY, Archambault P, English SW, Muscedere J, Serri K, Tarride JE, Mehta S, Verceles AC, Reeve B, O'Grady H, Kelly L, Strong G, Hurd AH, Thabane L, Cook DJ; CYCLE Investigators and the Canadian Critical Care Trials Group. Critical Care Cycling to Improve Lower Extremity Strength (CYCLE): protocol for an international, multicentre randomised clinical trial of early in-bed cycling for mechanically ventilated patients. BMJ Open. 2023 Jun 23;13(6):e075685. doi: 10.1136/bmjopen-2023-075685. PMID 37355270
- [Derived] Heels-Ansdell D, Kelly L, O'Grady HK, Farley C, Reid JC, Berney S, Pastva AM, Burns KE, D'Aragon F, Herridge MS, Seely A, Rudkowski J, Rochwerg B, Fox-Robichaud A, Ball I, Lamontagne F, Duan EH, Tsang J, Archambault PM, Verceles AC, Muscedere J, Mehta S, English SW, Karachi T, Serri K, Reeve B, Thabane L, Cook D, Kho ME. Early In-Bed Cycle Ergometry With Critically Ill, Mechanically Ventilated Patients: Statistical Analysis Plan for CYCLE (Critical Care Cycling to Improve Lower Extremity Strength), an International, Multicenter, Randomized Clinical Trial. JMIR Res Protoc. 2024 Oct 28;13:e54451. doi: 10.2196/54451. PMID 39467285
- [Derived] Kho ME, Berney S, Pastva AM, Kelly L, Reid JC, Burns KEA, Seely AJ, D'Aragon F, Rochwerg B, Ball I, Fox-Robichaud AE, Karachi T, Lamontagne F, Archambault PM, Tsang JL, Duan EH, Muscedere J, Verceles AC, Serri K, English SW, Reeve BK, Mehta S, Rudkowski JC, Heels-Ansdell D, O'Grady HK, Strong G, Obrovac K, Ajami D, Camposilvan L, Tarride JE, Thabane L, Herridge MS, Cook DJ. Early In-Bed Cycle Ergometry in Mechanically Ventilated Patients. NEJM Evid. 2024 Jul;3(7):EVIDoa2400137. doi: 10.1056/EVIDoa2400137. Epub 2024 Jun 12. PMID 38865147

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03471247/SAP_000.pdf